CLINICAL TRIAL: NCT03055351
Title: Stop&Go: an Intervention Program to Promote Healthy and Physically Active Lifestyles Among Patients With Substance Use Disorders
Brief Title: Stop&Go: an Intervention Program to Promote Healthy and Active Lifestyles Among Patients With Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-STO-2016-80
Record Dates: First submitted 2017-01-25; First posted 2017-02-16 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Substance Use Disorder; Motivation
Keywords: Exercise motivation; Psychological well-being; Healthy living; Physical activity; Autonomy support; Self-determination theory
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants will complete the outcome measures but will not receive any intervention.
- Stop&Go Intervention (Experimental): Participants in this group will participate in an intervention aimed at promoting a healthy and physically active lifestyle. The intervention will be based on Self-determination theory postulates and will have two axes: training and motivation.
  Interventions: Behavioral: Stop&Go Intervention

INTERVENTIONS:
Behavioral: Stop&Go Intervention — Stop&Go intervention will be based on Self-determination theory. Patients will participate in four practically-oriented training sessions, focused on (1) nutrition and oral hygiene, (2) sleep habits and self-care, (3) physical activity and exercise, and (4) smoking cessation. In addition, the entire inpatient detoxification centre will be adapted to encourage autonomous physical activity and to reinforce the ideas presented in the training sessions.
  Arms: Stop&Go Intervention

SUMMARY:
Stop&Go is an intervention program aimed at promoting a healthy and physically active lifestyle for patients requiring inpatient detoxification treatment. The program includes two different phases. Phase I is aimed at understanding the variables related with adherence to healthy lifestyle interventions. Phase II will use the knowledge obtained in Phase I to develop and evaluate an intervention based on Self-determination theory to promote healthy and physically active lifestyles for patients admitted to an inpatient detoxification centre. The Stop&Go intervention is hypothesized to help patients move towards a healthy lifestyle and thus, may bring about changes in patients' (1) knowledge acquired, (2) indicators of healthy habits (e.g., exercise motivation) and (3) psychological well-being and ill-being.

DETAILED DESCRIPTION:
In patients with substance use disorders, exercise could help in the treatment of substance addictions. Interventions focused on promoting physical activity and healthy lifestyle for patients in residential treatment centres and ambulatory settings have been developed in the last years. However, there is a lack of programs promoting a healthy and physically active lifestyle for patients requiring inpatient detoxification treatment. Thus, the plan is to develop an intervention program with such characteristics, namely "Stop&Go".

Stop&Go includes two different phases. Phase I is aimed at understanding the variables related with adherence to healthy lifestyle interventions. Patients with substance use disorders will be invited to participate in focus groups (Study 1) and to respond to questionnaires (Study 2) assessing variables related to exercise and healthy habits (e.g., intention to be physically active). Phase II will use the knowledge obtained in Phase I to develop and evaluate an intervention to promote healthy and physically active lifestyle for patients admitted to an inpatient detoxification centre. The intervention will be based on Self-determination theory postulates and will have two axes: to educate and to motivate. Patients will participate in four practically-oriented training sessions, focused on (1) nutrition and oral hygiene, (2) sleep habits and self-care, (3) physical activity and exercise, and (4) smoking cessation. In addition, the entire inpatient detoxification centre will be adapted to encourage autonomous physical activity and to reinforce the ideas presented in the training sessions.

The main strength of Stop&Go is expected to be the combination of perspectives included in its development (i.e., intervention led by an interdisciplinary team and based on patients' needs). The Stop&Go intervention is hypothesized to help patients move towards a healthy lifestyle and thus, may bring about changes in patients' (1) knowledge acquired, (2) variables related to healthy habits (e.g., exercise motivation) and (3) psychological well-being and ill-being.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-V criteria for substance use disorder.
* Request for treatment primarily based on substance detoxification.
* Voluntary admission to an impatient detoxification centre
* Age ≥ 18 years old.

Exclusion Criteria:

* Mental disorders that could hinder patient assessment
* Difficulty to answer the survey due to limited literacy or poor Spanish language proficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Changes from patients' baseline exercise motivations at the moment of discharge, measured with the Behavioural Regulation in Exercise Questionnaire (BREQ-3; Wilson et al., 2006). | Immediately upon admission to the centre, as well as upon successful discharge, measured up to a total of 10 days.
  The BREQ-3 measures 6 different types of exercise regulations: intrinsic motivation, integrated reg., identified reg., introjected reg., external reg., amotivation.
  Participants will be included in the study as they begin their inpatient detoxification treatment and will finish their participation when they are successfully discharged from the centre. Exercise motivations will be measured at 2 time points (Time 1- patient's admission to the detoxification centre, Time 2- successful discharge from the centre), but is not possible to specify in advance the exact number of days between time points due to the following main reason: This study is conducted in an inpatient detoxification unit and consequently medical criteria will prevail in order to estimate the varying duration of treatments. In any case, according to the best clinical practice, detoxification treatments usually last 11-15 days and thus it is expected that at least 10 days elapse between the aforementioned 2 time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No